CLINICAL TRIAL: NCT07284498
Title: Treatment of Seizures in Neonate With Hypoxic Ischemic Encephalopathy
Brief Title: Treatment of Seizures in Neonate With HIE
Acronym: HIE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdulwahab Uosef Alqarni, M.Sc, Mansoura University, PhD student, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDP.25.01.179
Record Dates: First submitted 2025-11-16; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Seizures; HIE - Hypoxic - Ischemic Encephalopathy
Keywords: Neonatal Seizure; HIE; Phenobarbital; Levetiracetam
MeSH Terms: interventions — Phenobarbital; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phenobarbital Arm ( Group A ) (Active Comparator): Patients in Group A will receive PHENobarbital at a loading dose of 20 mg/kg within a 20-minute time frame from the start of treatment. If the seizure dose is not stopped after 20 minutes, another 20 mg/kg of the same medication will be added, and if the seizure dose is not stopped within the total time frame of 40 minutes, this will be considered a treatment failure. If seizures are controlled, patients will receive a maintenance dose of PHENobarbital 3-5 mg/kg/day IV/PO, in 1-2 divided doses, starting 12 hours after the loading dose.
  Interventions: Drug: Phenobarbital
- Levetiracetam Standard Dose Arm ( Group B ) (Active Comparator): Patients in Group B will receive levETIRAcetam at a loading dose of 30 mg/kg within a timeframe of 20 minutes from the start of seizures if the seizures don't stop. The same beginning dose will be repeated, in case the seizures don't stop within the 40-minute time frame, which leads to the treatment being considered a failure and a need to move to the second line of treatment. If seizures are controlled, patients will receive maintenance dose of levETIRAcetam 30 mg/kg/day IV or orally, divided into three daily doses.
  Interventions: Drug: Levetiracetam
- Levetiracetam High Dose Arm ( Group C ) (Active Comparator): Patients in Group C will receive levETIRAcetam at a loading dose of 60 mg/kg within a timeframe of 20 minutes from the start of seizures if the seizures don't stop. The same beginning dose will be repeated, in case the seizures don't stop within the 40-minute time frame, which leads to the treatment being considered a failure and a need to move to the second line of treatment. If seizures are controlled, patients will receive maintenance dose of levETIRAcetam 60 mg/kg/day IV or orally, divided into three daily doses.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Phenobarbital — Phenobarbital is strongly recommended by the World Health Organization as the first-line treatment of neonatal seizures and is the standard of care at most institutions
  Arms: Phenobarbital Arm ( Group A )
Drug: Levetiracetam — levetiracetam has emerged as an alternative Anti-seizure medication that may offer improved safety and tolerability profiles.
  Arms: Levetiracetam High Dose Arm ( Group C ); Levetiracetam Standard Dose Arm ( Group B )

SUMMARY:
Aim of the study To evaluate and compare phenobarbital's and levetiracetam's safety and efficacy for treating seizures in neonates with moderate to severe HIE

DETAILED DESCRIPTION:
This research will be conducted as a randomized controlled open-labeled single-centered clinical trial. The Declaration of Helsinki will guide the study's conduct. Informed consents will be obtained from neonates' parents, and the local ethical committee approval is mandatory.

Baseline data as detailed medical history, physical examination, gestational age, postnatal age, birth weight, APGAR score at 5 and 10 minutes. Laboratory parameter (complete blood cell count, electrolytes, serum creatinine, liver enzymes, and blood gas), respiratory assessment (need for oxygen and respiratory support), cardiac assessment including (blood pressure/ heart rate), type of feeding, head ultrasound.

The enrolled patients will be classified into three groups: Phenobarbital group (intervention group A), Levetiracetam standard dose group (intervention group B), Levetiracetam high dose group (intervention group C).

Patients in Group A (intervention group I) will receive phenobarbital at a loading dose of 20 mg/kg within a 20-minute time frame from the start of seizures. If the seizures doesn't stopped after 20 minutes, another 20 mg/kg of the same medication will be added, and if the seizures doesn't stopped within the total time frame of 40 minutes, this will be considered a treatment failure.

While patients in Group B (Intervention Group II) as well as Group C (Control Group) will receive levetiracetam at a loading dose of 30 mg/kg and 60 mg/kg respectively. Within a timeframe of 20 minutes from the start of seizures, If the seizures doesn't stopped. The same beginning dose will be repeated for both groups, in case of seizures doesn't stopped within the 40-minute time frame, which leads to the treatment being considered a failure and a need to move to the second line of treatment.

For all groups, if the first line of treatment fails, phenytoin will be considered as the second line treatment for treating seizures, and a dose of (20 mg/kg diluted in 20 ml of saline solution over 20 minutes) will be started. If the seizures is not controlled, the third line will be midazolam, given as a continuous infusion.

Evaluations will include patients who will be followed up during the study period by measuring the following parameters: frequent episodes of seizure/ time to stop seizures, EEG finding, follow-up head ultrasound (US) and brain magnetic resonance imaging (MRI) (if the neonate-stable), blood pressure/ heart rate (need for inotrope/vasopressor treatment), respiratory status (need for oxygen and respiratory support), feeding intolerance (vomiting); and changes in laboratory parameters (complete blood cell count to assess anemia, electrolytes, serum creatinine, liver enzymes, ammonia, and arterial blood gas (ABG) analysis or any significant side effects that were attributed to an anti-seizures medication by the clinical team and will be recorded in the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates diagnosed with moderate or severe HIE.
2. Presence of clinical seizures (focal / generalized tonic /colonic, myoclonic, subtle and spasms) and/or documented amplitude electroencephalogram (aEEG) abnormality within the first 72 hours.

Exclusion Criteria:

1. Exclusive metabolic causes.
2. Serum creatinine greater than 1.6 mg/dl.
3. Known pyridoxine-dependent seizures.
4. Prior treatment with anti-epileptic drugs.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of findings anti-seizure Medication safety and efficacy | 24-hour seizure-free period.
  A complete 24-hour seizure-free period is measured and assessed by clinical symptoms and/or an independent aEEG assessment of seizure-free within 20 to 40 minutes of initiating drug therapy, without the need for second-line antiepileptic therapy.

SECONDARY OUTCOMES:
Comparison of the effectiveness of anti-seizure medications for 48 continuous hours after the start of treatment. | 48 hours after initiation of treatment
  1. Sustained seizure cessation (48 h):
     Absence of clinical or electrographic seizures for ≥48 consecutive hours after antiseizure therapy.
     Unit: Yes/No
  2. Need for inotropes/vasopressors:
     Requirement for vasoactive agents (e.g., dopamine) for hypotension within 48 hours.
     Unit: Yes/No
  3. Respiratory support requirement: Need for supplemental oxygen or ventilatory support (CPAP/NIV/mechanical ventilation).
     Unit: Yes/No
  4. Feeding intolerance:
     Vomiting, abdominal distension, or interruption of enteral feeding. Unit: Yes/No
  5. Hematologic abnormalities:
     Anemia (Hb <13 g/dL), thrombocytopenia (platelets <150×10⁹/L), or leukopenia (WBC <5×10⁹/L).
     Unit: ×10³/µL
  6. Electrolyte disturbances:
     Abnormal Na, K, Ca, or glucose levels per neonatal reference ranges. Unit: mmol/L
  7. Acute liver injury:
     AST or ALT >2× age-adjusted upper limit. Unit: IU/L
  8. Hyperammonemia:
     Plasma ammonia >100 µmol/L. Unit: µmol/L
  9. Abnormal blood gas:
  Metabolic or respiratory acidosis: pH <7.25 and/or BE ≤ -10 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Moetaza Soliman, Associate Professor, Principal Investigator — Faculty of Pharmacy, Mansoura University; Nada Abdelfattah, Associate Professor, Principal Investigator — University Children's Hospital, Mansoura University
Locations (2):
- Egypt (2):
  - University Children's Hospital, Mansoura University, Al Mansurah
  - Al Galaa Teaching Hospital, Cairo

REFERENCES:
- [Result] Finster M, Wood M. The Apgar score has survived the test of time. Anesthesiology. 2005 Apr;102(4):855-7. doi: 10.1097/00000542-200504000-00022. PMID 15791116
- [Result] Sarnat HB, Sarnat MS. Neonatal encephalopathy following fetal distress. A clinical and electroencephalographic study. Arch Neurol. 1976 Oct;33(10):696-705. doi: 10.1001/archneur.1976.00500100030012. PMID 987769
- [Result] Susnerwala S, Joshi A, Deshmukh L, Londhe A. Levetiracetam or Phenobarbitone as a First-Line Anticonvulsant in Asphyxiated Term Newborns? An Open-Label, Single-Center, Randomized, Controlled, Pragmatic Trial. Hosp Pediatr. 2022 Jul 1;12(7):647-653. doi: 10.1542/hpeds.2021-006415. PMID 35673948
- [Result] Qiao MY, Cui HT, Zhao LZ, Miao JK, Chen QX. Efficacy and Safety of Levetiracetam vs. Phenobarbital for Neonatal Seizures: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Nov 18;12:747745. doi: 10.3389/fneur.2021.747745. eCollection 2021. PMID 34867732
- [Result] Gyandeep G, Behura SS, Sahu SK, Panda SK. Comparison between Phenobarbitone and Levetiracetam as the initial anticonvulsant in preterm neonatal seizures - a pilot randomized control trial in developing country setup. Eur J Pediatr. 2023 May;182(5):2133-2138. doi: 10.1007/s00431-023-04864-x. Epub 2023 Feb 24. PMID 36823477
- [Result] Verwoerd C, Limjoco J, Rajamanickam V, Knox A. Efficacy of Levetiracetam and Phenobarbital as First-Line Treatment for Neonatal Seizures. J Child Neurol. 2022 Apr;37(5):401-409. doi: 10.1177/08830738221086107. Epub 2022 Mar 20. PMID 35311411
- [Result] Efficacy of levetiracetam as the first line anti- epileptic drug in management of neonatal seizures
- [Result] Battig L, Dunner C, Cserpan D, Ruegger A, Hagmann C, Schmitt B, Pisani F, Ramantani G. Levetiracetam versus Phenobarbital for Neonatal Seizures: A Retrospective Cohort Study. Pediatr Neurol. 2023 Jan;138:62-70. doi: 10.1016/j.pediatrneurol.2022.10.004. Epub 2022 Oct 22. PMID 36401982
- [Result] Sharpe C, Reiner GE, Davis SL, Nespeca M, Gold JJ, Rasmussen M, Kuperman R, Harbert MJ, Michelson D, Joe P, Wang S, Rismanchi N, Le NM, Mower A, Kim J, Battin MR, Lane B, Honold J, Knodel E, Arnell K, Bridge R, Lee L, Ernstrom K, Raman R, Haas RH; NEOLEV2 INVESTIGATORS. Levetiracetam Versus Phenobarbital for Neonatal Seizures: A Randomized Controlled Trial. Pediatrics. 2020 Jun;145(6):e20193182. doi: 10.1542/peds.2019-3182. Epub 2020 May 8. PMID 32385134
- [Result] Hooper RG, Ramaswamy VV, Wahid RM, Satodia P, Bhulani A. Levetiracetam as the first-line treatment for neonatal seizures: a systematic review and meta-analysis. Dev Med Child Neurol. 2021 Nov;63(11):1283-1293. doi: 10.1111/dmcn.14943. Epub 2021 Jun 13. PMID 34124790
- [Result] Akeel NE, Suliman HA, Al-Shokary AH, Ibrahim AO, Kamal NM, Abdelgalil AA, Elmala MK, Elshorbagy HH, Nasef KA, Attia AM, Fathallah MGED. A Comparative Study of Levetiracetam and Phenobarbital for Neonatal Seizures as a First Line Treatment. Glob Pediatr Health. 2022 Dec 20;9:2333794X221143572. doi: 10.1177/2333794X221143572. eCollection 2022. PMID 36578326